CLINICAL TRIAL: NCT00561522
Title: Capecitabine as Adjuvant Chemotherapy to Prevent Recurrence of Hepatocellular Carcinoma After Curative Resection: a Randomized Controlled Trial
Brief Title: Capecitabine to Prevent Recurrence of Hepatocellular Carcinoma After Curative Resection
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Zhongshan Hospital, Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-07-RCT-LCI1
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2010-07-21 (Estimated); Status verified 2009-08

CONDITIONS: Hepatocellular Carcinoma; Neoplasm Metastasis
Keywords: Recurrence; Metastasis; Hepatocellular Carcinoma; Radical Hepatic Resection; Drug Prevention; Capecitabine; Surgery
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasm Metastasis; Recurrence | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention treatment (Experimental): Capecitabine
  Interventions: Drug: Capecitabine
- No intervention treatment (No Intervention): No other preventive treatment
  Interventions: Other: No other preventive treatment

INTERVENTIONS:
Drug: Capecitabine — Capecitabine 1,250 mg/m2 twice daily on days 1-14, followed by a 7-day drug-free interval. Treatment repeats every 21 days. The above cycle is repeated for 4-6 times.If disease recurrence or unacceptable toxicity or other criteria for withdrawal are met, treatment will be stopped.
  Arms: Intervention treatment
Other: No other preventive treatment — No other preventive treatment
  Arms: No intervention treatment

SUMMARY:
The purpose of this study is to determine whether capecitabine is effective to prevent disease recurrence after curative hepatic resection in patients with hepatocellular carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) accounts for 70-90% of primary liver cancers, which is the third most common cause of death from cancer worldwide; over half a million new cases are diagnosed worldwide each year. Hepatic resection has been established as one of the most effective and safe therapeutic options for HCC. However, recurrence, particularly metastatic recurrence, is one of the major obstacles to long-term survival. Several adjuvant treatments have been used to prevent recurrence after surgery, but their effectiveness remains controversial. Fluorouracil (FU), an antimetabolite, is a commonly used chemotherapeutic agent, with activity in a variety of solid tumors including those of the head and neck, breast, prostate, pancreas, liver, and genitourinary and gastrointestinal tracts. Capecitabine (Xeloda; Roche), a novel prodrug of 5-FU, is an orally administered tumor-selective cytotoxic agent that is converted to 5-FU by three enzymes. Capecitabine has the advantages of convenient oral administration and of mimicking the effect of protracted intravenous (i.v.) 5-FU. Capecitabine is currently approved by the FDA for use as first-line therapy in patients with metastatic colorectal cancer when single-agent fluoropyrimidine therapy is preferred. The drug is also approved for use as a single agent in metastatic breast cancer patients who are resistant to both anthracycline- and paclitaxel-based regimens or in whom further anthracycline treatment is contraindicated. Our previous study found that PD-ECGF mRNA was highly expressed in human HCC and particularly in portal vein tumor thrombus as compared with noncancerous liver tissues. Capecitabine inhibits tumor growth and metastatic recurrence after resection of HCC in highly metastatic nude mice model. The effect of capecitabine may be attributed to the high expression of PD-ECGF in tumors. The antitumor activity of single-agent capecitabine was modest in patients with HCC, including those with cirrhosis. Von Delius et al reported that capecitabine was found to be safe for treatment of patients with HCC, including those with compensated cirrhosis. On the basis of previous findings, we designed a randomized, controlled trial to test the hypothesis that adjuvant postoperative chemotherapy with capecitabine can prevent tumor recurrence after radical hepatic resection in patients with HCC. Because capecitabine is administered orally, we considered that this treatment would be clinically useful if its effectiveness could be confirmed.

ELIGIBILITY:
Inclusion Criteria:

* First curative hepatic resection
* Hepatocellular Carcinoma (histologically confirmed)
* Cirrhosis of Child-Pugh class A or B
* A performance status ≤ 2
* Adequate bone marrow ,hepatic and renal functions (white blood cell (WBC) count > 2.5×10^3/μL, platelet count > 40×10^3/μL, a serum bilirubin level, alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 2 times the upper limit of the normal value, and serum creatinine level < 1.5 mg/dL)
* Major organ (heart, lung and brain) function was normal
* An age between 18 and 79 years.

Exclusion Criteria:

* Any active infectious process
* Known hypersensitivity to capecitabine
* The presence of clinically confirmed extrahepatic metastasis, macroscopic evidence of tumor thrombus in the inferior vena cava or the main portal vein or the main bile duct
* Other previous or synchronous malignant disorders
* Postoperative dysfunction of any organ.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2007-11; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
The primary end point was to determine the effect on disease-free survival and overall survival by oral capecitabine. | four years

SECONDARY OUTCOMES:
The secondary end point was to analyze the relationship between preventive effectiveness of capecitabine with thymidine phosphorylase expression level of tumor tissue. | four years

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, M.D., Study Director — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China